CLINICAL TRIAL: NCT05801718
Title: Growth Parameters & Body Mass Index in Children With Chronic Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Norhan Nabil Ahmed, resident at pediatric department at Sohag university hospital, Sohag University
Other Study IDs: Soh-Med-23-03-09MS
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Chronic Medical Diseases
MeSH Terms: interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- chronic cardiac patients: patients with chronic cardiac diseases affecting their groth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic renal patients: patients with chronic renal diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic respiratory diseases: patients with chronic respiratory diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic metabolic diseases: patients with chronic metabolic diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic neurological diseases: patients with chronic neurological diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic haematological diseases: patients with chronic haematological diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index
- chronic gastro-intestinal diseases: patients with chronic gastro-intestinal diseases affecting their growth parameters & body mass index
  Interventions: Diagnostic Test: Growth parameters & body mass index

INTERVENTIONS:
Diagnostic Test: Growth parameters & body mass index — measuring the anthropometric measurements including: Weight, height/ length, head circumference, mid arm circumference& skin fold thickness and measuring body mass index.

SUMMARY:
Deviations from the normal pattern of growth may be the first clues to pathology as in many chronic diseases evaluated clinically by anthropometric measurements & body mass index. Growth impairment in children with chronic diseases is associated with disruption of the growth hormone (GH) and predominantly results from undernutrition, chronic inflammation and prolonged corticosteroid treatment.

Undernutrition leads to major adaptations in the endocrine system towards conserving energy, diverting substrates away from growth and reproduction, and providing alternative sources of energy for critical body homeostasis. chronic inflammatory processes exacerbate undernutrition through proinflammatory cytokines such as interleukin-1&6 and tumor necrosis factor. These growth-regulating mechanisms are disturbed further by corticosteroids used in some chronic conditions for their anti-inflammatory and immunosuppressive properties.

Growth impairment occurs with many chronic conditions e g: Congenital heart dieases (CHD), chronic pulmonary diseases such as bronchial asthma, Gastrointestinal diseases sch as inflammatory bowel disease ,Chronic liver diseases , Chronic renal diseases, Chronic hemolytic anemia and chronic Central nervous system diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age: under 12 years old.
* Both sex .
* Patients with chronic medical diseases.

Exclusion Criteria:

* Age: over 12years old.
* Patients with acute diseases.
* Pediatric with malignancy.
* chronic patients with surgical sequelae.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children with chronic diseases affecting their growth parameters & body mass index.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Weight | one year
  For children less than two years of age, use a calibrated beam or a digital infant scale. Ensure the infant is not wearing any clothes and remove the diaper before measuring the weight. The weight should be measured to the nearest 0.01 kg or 0.5 ounces. For children older than 24 months, a balanced floor scale or electronic floor scale can be used.
Height | one year
  For children who can stand, a stadiometer should be used. The child should stand up straight, with buttocks, shoulder blades, and heels together touching the back of the stadiometer. The feet should face outward at a 60-degree angle. If the patient has genu valgum, separate the feet enough to avoid overlapping the knees while maintaining contact between the knees. Arms should be loosely hanging at the sides with palms facing the thighs. The horizontal bar of the stadiometer should be lowered until the hair is compressed to the crown of the head. Remove any objects on the head and hair that may obstruct the bar from compressing the hair to the crown of the head. The measurement should be read to the nearest 0.1 cm or 1/8 of an inch. Repeat the measurement twice to obtain two readings within 0.2cm or 0.25 inches. The average of the two closest measurements should be recorded.
Length | one year
  For infants and toddlers who cannot stand, the recumbent length should be measured. Align the infant's head against the top of the headboard of the infantometer. An assistant must straighten the infant's body and legs, ensuring the feet are parallel to the footboard. Repeat the measurement twice to obtain two readings within 0.2 cm or 0.25 inches. The average of the two closest measurements should be recorded.
Head circumference | one year
  For infants and toddlers less than two years of age, measure the largest circumference of the head using a non-stretchable measuring tape around the most prominent part of the head to the middle of the forehead. The tape measure should be pulled snug around the head to compress the hair and underlying soft tissue. Repeat the measurement twice to obtain two readings within 0.2 cm or 0.25 inches. The average of the two closest measurements should be recorded.
Mid arm circumference | one year
  The patient stands upright with the arm hanging freely at the side. The patient should not flex the arm muscles. Measuring tape should be placed snugly around the mid-point of the arm without compressing the skin.
Skin fold thickness | one year
  Common sites for skinfold measurements include the biceps, triceps, iliac crest, thigh, calf, subscapular, abdomen, and chest. The exact technique can vary, but we will discuss one method using the triceps as an example. For the triceps skinfold, grab the skin 2 cm above the midpoint of the right upper arm with the thumb and index finger to create a skinfold. Then, place the calipers at the midpoint to obtain the measurement. Similarly, at other sites, the skinfold measurement is obtained by grabbing the skin 2 cm away from the measuring site. Despite standard measuring techniques, skinfold testing has high variability and has limited use thus far in the clinical setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costello CL, Gellatly M, Daniel J, Justo RN, Weir K. Growth Restriction in Infants and Young Children with Congenital Heart Disease. Congenit Heart Dis. 2015 Sep-Oct;10(5):447-56. doi: 10.1111/chd.12231. Epub 2014 Nov 11. PMID 25385245
- [Background] Rodig NM, McDermott KC, Schneider MF, Hotchkiss HM, Yadin O, Seikaly MG, Furth SL, Warady BA. Growth in children with chronic kidney disease: a report from the Chronic Kidney Disease in Children Study. Pediatr Nephrol. 2014 Oct;29(10):1987-95. doi: 10.1007/s00467-014-2812-9. Epub 2014 Apr 12. PMID 24728472
- [Background] Amaro F, Chiarelli F. Growth and Puberty in Children with Inflammatory Bowel Diseases. Biomedicines. 2020 Oct 29;8(11):458. doi: 10.3390/biomedicines8110458. PMID 33138015
- [Background] Hauspie R, Susanne C, Alexander F. Maturational delay and temporal growth retardation in asthmatic boys. J Allergy Clin Immunol. 1977 Mar;59(3):200-6. doi: 10.1016/0091-6749(77)90150-6. PMID 190283